CLINICAL TRIAL: NCT01622049
Title: Selective Laser Photocoagulation of Communicating Vessels in Twin-Twin Transfusion Syndrome
Acronym: TTTS
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: #105118
Record Dates: First submitted 2010-08-05; First posted 2012-06-18 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2012-11

CONDITIONS: Twin Twin Transfusion Syndrome
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TTTS treatment method: This is an observational trial. Patients who meet eligibility criteria and give written informed consent will have SLPCV. All subjects will receive ongoing standard-of-care prenatal care for the duration of their pregnancy from their referring perinatologist or obstetrician.
  Interventions: Device: Selective Laser Photocoagulation of Communicating Vessels

INTERVENTIONS:
Device: Selective Laser Photocoagulation of Communicating Vessels — Patients will be admitted to Tampa General Hospital. Laboratory tests and anesthesia assessments will be completed. Antibiotic prophylaxis is initiated within an hour of surgery and continued every 8 hours through the first post-operative day. Surgery will be performed preferably under local anesthesia for the mother using 1% xylocaine with epinephrine at the trocar entry site, and IV sedation. Surgery will be performed with standard operative fetoscopy equipment and techniques. A trocar will be introduced in the amniotic cavity of the recipient. An amniotic fluid sample will be obtained for microbiological studies, and genetic analysis for clinical care only. The amniotic fluid will be discarded after analysis. The communicating vessels will be located endoscopically and will be lasered with YAG laser energy. The procedure will be monitored both endoscopically and sonographically. The presence of fetal heart activity will be noted. An amniodrainage of the larger sac may be performed
  Other Names: SLPCV

SUMMARY:
Patients undergo a detailed ultrasound examination to rule out the presence of congenital anomalies, and to assess the hemodynamic status of the fetuses. Patients with confirmed TTTS will be considered candidates for the trial. Patients will be counseled about the risks and benefits of all treatment options and will be free to choose any treatment option. They will then be asked to sign an informed consent. The procedure will be performed under local anesthesia. After a 2-3 mm skin incision, and under ultrasound guidance, the trocar will be introduced in the amniotic cavity of the Recipient twin. The communicating vessels will be located endoscopically and will be lasered with YAG laser energy. An accessory port may be required in some cases. The procedure will be monitored both endoscopically and sonographically. The presence of fetal heart activity will be noted often during the procedure. An amniodrainage of the larger sac may be performed at the time of the procedure. The patient will remain hospitalized 1-3 days and will undergo an ultrasound assessment on the first post operative day. Patients will undergo a weekly ultrasound examination for four weeks after the initial therapeutic procedure. Sonographic parameters to evaluate will include: maximum vertical pocket of fluid in each sac, visualization of the fetal bladders, absence or presence of hydrops, and Doppler studies of the umbilical artery, umbilical vein, ductus venosus, and middle cerebral artery. After delivery babies will be assessed by their corresponding neonatologists or pediatricians. Infants admitted to the neonatal intensive care unit will be followed through their discharge. Evidence of neurological or cardiac morbidity will be sought in each twin. If either of these complications is suspected, evaluation by pediatric neurology or pediatric cardiology will be requested. Babies will be followed up for neonatal, infant and childhood morbidity or mortality. It is requested that all placentas be delivered fresh to Tampa General Hospital in an icebox container for assessment. Placentas will be discarded after analysis.

ELIGIBILITY:
Inclusion Criteria

To be eligible, patients must meet the following criteria:

1. Maternal age 18 to 55 years
2. Gestational age: 16 weeks, 0 days to 26 weeks, 0 days.
3. Confirmed TTTS patients, who by definition meet the following sonographic criteria:

   1. Single placenta.
   2. Polyhydramnios: maximum vertical pocket >= 8 cm in the recipient twin, prior to amniodrainage.
   3. Oligohydramnios: maximum vertical pocket <=2 cm in the donor twin, prior to amniodrainage.
   4. Thin dividing membrane (absence of twin peak sign) or absence of dividing membrane (monoamniotic).
   5. Same gender, if visible.
4. Patients choosing laser therapy that have undergone prior therapeutic amniocentesis may be included.
5. Patients with an anterior placenta may be included.
6. Triplet gestations with two or three fetuses sharing the same placenta may be included.
7. Patients must be able to give written informed consent. Inclusion Criteria 5.2 Exclusion Criteria

The following criteria would exclude patients from participation in the study:

1. Patients unable or unwilling to participate in the study or to be followed up.
2. Patients unable to give written informed consent.
3. Presence of major congenital anomalies that may not warrant surgery.
4. Known unbalanced chromosomal complement.
5. Prior intentional septostomy (purposely making a hole in the dividing membrane).
6. Ruptured membranes.
7. Chorioamnionitis.
8. Abnormal intracranial ultrasound findings of either fetus to include, but not limited to: intraventricular hemorrhage, porencephalic cysts, hydrocephalus, Dandy-Walker syndrome, holoprosencephaly and agenesis of the corpus callosum. Isolated ventriculomegaly (atrium 10-19 mm) may or may not be used an exclusion criteria.
9. Placental abruption.
10. Active labor.
11. Jehovah's Witness.
12. Any other patient deemed inappropriate for the study by the principal investigator.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2006-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to evaluate neonatal/infant survival 6 months after birth. | 6 months

SECONDARY OUTCOMES:
The secondary study objective is to evaluate the effects of surgery on postnatal neurological morbidity. For the purposes of this clinical trial, neurological morbidity includes any of the following conditions diagnosed within 6 months of birth | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A Quintero, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

REFERENCES:
- [Result] Chmait RH, Kontopoulos EV, Korst LM, Llanes A, Petisco I, Quintero RA. Stage-based outcomes of 682 consecutive cases of twin-twin transfusion syndrome treated with laser surgery: the USFetus experience. Am J Obstet Gynecol. 2011 May;204(5):393.e1-6. doi: 10.1016/j.ajog.2011.02.001. Epub 2011 Mar 15. PMID 21411051